CLINICAL TRIAL: NCT07299955
Title: A Phase 1, Randomized, Double-Blind, Two-arm, Parallel Design, Comparative Study to Assess Pharmacokinetics, Immunogenicity, Safety and Tolerability of Bmab3000 and Herceptin Hylecta® Following a Single Dose of 600 mg Subcutaneous Injection in Healthy Male Volunteers
Brief Title: A Phase 1 Comparative Study to Evaluate Pharmacokinetics, Immunogenicity, Safety and Tolerability of Bmab3000 and Herceptin Hylecta® After a Single 600 mg SC Injection in Healthy Male Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biocon Biologics UK PLC (Industry)
Responsible Party: Sponsor
Organization: Biocon Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-TRASTU-103; U1111-1329-7865 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy Male Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bmab3000 (Experimental): Single s.c. dose of Bmab3000 containing 600 mg of trastuzumab and 10,000 units of hyaluronidase in 5 mL
  Interventions: Biological: Herceptin Hylecta®
- Herceptin Hylecta® (Active Comparator): Single s.c. dose of Herceptin Hylecta containing 600 mg of trastuzumab and 10,000 units of hyaluronidase in 5 mL
  Interventions: Biological: Bmab3000

INTERVENTIONS:
Biological: Bmab3000 — Single s.c. dose of Bmab3000 containing 600 mg of trastuzumab and 10,000 units of hyaluronidase in 5 mL
  Arms: Herceptin Hylecta®
Biological: Herceptin Hylecta® — Single s.c. dose of Herceptin Hylecta containing 600 mg of trastuzumab and 10,000 units of hyaluronidase in 5 mL
  Arms: Bmab3000

SUMMARY:
This phase I study is to compare the pharmacokinetics (PK), immunogenicity, safety, and tolerability of Bmab3000 (test) and Herceptin Hylecta (reference) after a single subcutaneous (s.c.) dose in healthy male volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, two-arm, parallel-group trial comparing the pharmacokinetics (PK), immunogenicity, safety, and tolerability of Bmab3000 (test) and Herceptin Hylecta (reference) after a single subcutaneous (s.c.) dose.

A total of 150 healthy male participants (75 per arm) will be enrolled to ensure 138 evaluable subjects. Participants will be randomized in 1:1 using stratified block randomization based on baseline body weight (≥50-≤75 kg and >75-≤100 kg).

Each participant will be involved in the study for approximately four months, which includes one screening visit, a 3-night inpatient stay, and 16 scheduled outpatient follow-up visits. Participants will attend a screening visit (Day -28 to Day -1) to confirm eligibility. This will include obtaining informed consent, medical history, physical examination, vital signs, biometric measurements, ECG, echocardiogram, and blood and urine tests, as well as drug and alcohol screening. Eligible participants will be admitted to the study site on Day -1 for pre-dose assessments to confirm continued eligibility. On Day 1, participants will receive a single subcutaneous injection of either Bmab3000 or Herceptin Hylecta. During the inpatient stay (Days -1 to 3), participants will undergo continuous safety monitoring, including regular vital signs, ECGs, injection site checks, and blood sampling for pharmacokinetic, safety, and immunogenicity assessments. After discharge, participants will return for outpatient visits till Day 85 for continued safety monitoring, blood sampling for pharmacokinetic and immunogenicity analyses, and ECGs and vital sign assessments. The final visit on Day 91 will include a full physical examination, echocardiogram, ECG and blood sampling for pharmacokinetic & immunogenicity analyses and final laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged between 18 to 65 years; both inclusive.
2. Body weight ≥50 kg and ≤100 kg with body mass index (BMI) between 18.5 and 30 kg/m2, both inclusive.
3. Participants should have Left ventricular ejection fraction (LVEF) ≥55%.
4. Male participants must be using an acceptable method of contraception for the entire duration of the trial, and for at least three months after the trial drug administration. Participants must refrain from fathering a child or donating sperm in the next three months following the last trial drug administration or undergoing vasectomy.
5. All non-prescription medications must have been discontinued at least 14 days prior to dosing.
6. All non-topical prescription medications must have been stopped at least 30 days prior to admission to the clinical research center.
7. Absence of significant findings in the vital signs, 12 lead ECG, and clinical laboratory tests of blood and urine.
8. Willing and able to sign the informed consent form (ICF).

Exclusion Criteria:

1. History of previous exposure to trastuzumab.
2. Presence of clinically significant medical history and clinically significant findings in the physical examination.
3. Allergy or hypersensitivity to trastuzumab, other recombinant human or humanized antibodies, other related products, or any excipients/ ingredients (e.g. hyaluronidase).
4. Sick sinus syndrome or known long QT syndrome (QTcF >450 msec).
5. Pronounced sinus bradycardia (<40 bpm), even if elicited by sport.
6. History of relevant drug and/or food allergies.
7. Positive urine drug and breath alcohol screen.
8. Consumption of any foods containing poppy seeds within 48 hours (2 days) prior to screening/admission to the clinical research center.
9. Positive screen for hepatitis B surface antigen (HBsAg), anti-hepatitis virus (HCV) antibodies, anti-human immunodeficiency virus (HIV) 1 and 2 antibodies.
10. Donation or loss of blood prior to drug administration.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male volunteers aged between 18 to 65 years; both inclusive.
Enrollment: 150 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1 to Day 91
  Maximum observed concentration (Cmax) of drug Bmab 3000
AUCo-∞ | Day 1 to Day 91
  Comparison of area under the concentration-time curve from time 0 to infinity (AUC0-inf)

SECONDARY OUTCOMES:
AUCo-t | Day 1 to Day 91
  Area Under the serum Concentration versus time curve from time 0 to the last sampling time at which concentrations were at or above the limit of quantification
Tmax | Day 1 to Day 91
  Time to maximum observed concentration
Vd/F | Day 1 to Day 91
  Volume of distribution
Cl/F | Day 1 to Day 91
  drug clearance
t1/2 | Day 1 to Day 91
  Apparent terminal elimination half-life
AUC% extrapolation | Day 1 to Day 91
  % of the AUC that has been derived after extrapolation
λz | Day 1 to Day 91
  Elimination rate constant

OTHER OUTCOMES:
Safety_ Adverse Reactions | Baseline to Day 91
  Adverse Events and Adverse Reactions during the Treatment Period
Safety_ Injection-site Reactions | Day 1 to Day 91
  Injection-site Reactions
Immunogenicity | Day 1 to Day 91
  Developing Antidrug Antibodies
Immunogenicity | Day 1 to Day 91
  Developing Neutralizing Antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Dr Cory Sellwood, MBBS, Principal Investigator — New Zealand Clinical Research (NZCR) Main Building: 264 Antigua Street, Christchurch, New Zealand; Dr Leanne Barnett, MBBS, Principal Investigator — New Zealand Clinical Research (NZCR) Main Building: 3 Ferncroft Street, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No